CLINICAL TRIAL: NCT02691026
Title: A Phase II Study of Pembrolizumab in Patients With Malignant Peripheral Nerve Sheath Tumor (MPNST), Not Eligible for Curative Surgery
Brief Title: A Study of Pembrolizumab in Patients With Malignant Peripheral Nerve Sheath Tumor (MPNST), Not Eligible for Curative Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment as a result of low incidence of MPNST and the COVID-19 pandemic.
Sponsor: Oslo University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Tormod Kyrre Guren, MD, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK3475_MPNST
Record Dates: First submitted 2016-02-04; First posted 2016-02-24 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Malignant Peripheral Nerve Sheath Tumour (MPNST)
Keywords: MPNST; Pembrolizumab
MeSH Terms: conditions — Neurofibrosarcoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pembrolizumab (Experimental): 200 mg pembrolizumab, i.v. infusion every 3 weeks for up to 10 cycles
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: Keytruda

SUMMARY:
This is phase II, single arm, open-label, interventional trial of pembrolizumab (MK-3475) in subjects with metastatic or locally advanced/unresectable or metastatic malignant peripheral nerve sheath tumour (MPNST).

The patients will be treated with pembrolizumab for up to 10 cycles.

Primary objective is to evaluate the percentage of patients with curatively unresectable MPNST who have achieved clinical response; complete response (CR), partial response (PR), or stable disease (SD) at 18 weeks as assessed by the Investigator, by using RECIST, v1.1.

DETAILED DESCRIPTION:
Patients with MPNST, who are not eligible for surgery of curative intent, will be considered for treatment with pembrolizumab. Patients will receive pembrolizumab treatment for up to 10 cycles. The patients must discontinue study treatment earlier (before 10 cycles of pembrolizumab) if they experience symptomatic deterioration attributed to disease progression, intolerable toxicity related to pembrolizumab, any medical condition that may jeopardize the patient's safety, use of other non-protocol anti-cancer therapy or pregnancy.

Patients who have received 10 cycles of pembrolizumab or discontinued study treatment of another reason than progression, will in the follow-up period be assessed for safety and treatment-related toxicity (for up to 90 days), progression and survival.

Patients who have achieved a clinical meaningful response after 10 cycles of pembrolizumab, defined as complete response (CR), partial response (PR), and stable disease (SD) assessed by the Investigator by using RECIST, v1.1, and have not experienced any clinically significant toxicity of study treatment, may be considered for reintroduction of pembrolizumab, if progression is detected after cycle 10.

Due to the low incidence of MPNST, the inclusion rate is expected to be low, thus a Simon's two-stage design is suggested (see Statistical Analysis Plans - Section 8.0).

Evaluation of efficacy and safety in stage one will be performed after the first 7 patient has been treated for 18 weeks: In case of no responders; the trial ends. If one or more responders, the trial will continue into stage two to a total number of 18 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have measurable disease based on RECIST, version 1.1.
4. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
5. Be willing to provide tissue from a newly obtained core or excisional biopsy of benign neurofibromatosis lesion (NF1 patients only)
6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
7. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least stable disease after 18 weeks of treatment assessed by RECIST 1.1. | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tormod K Guren, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo university Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No